CLINICAL TRIAL: NCT04672460
Title: A PHASE 1, OPEN LABEL, CROSSOVER STUDY TO ESTABLISH BIOEQUIVALENCE BETWEEN THE PROPOSED SOFT GEL TALAZOPARIB CAPSULE FORMULATION AND THE CURRENT TALAZOPARIB COMMERCIAL FORMULATION AND TO ESTIMATE THE FOOD EFFECT ON PHARMACOKINETICS OF THE PROPOSED TALAZOPARIB SOFT GEL CAPSULE FORMULATION IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: A Bioequivalence Study Between the Proposed and Current Talazoparib Capsule Formulation and Food Effect Study for the Proposed Talazoparib Capsule Formulation in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C3441037; 2020-006101-35 (EudraCT Number)
Record Dates: First submitted 2020-11-13; First posted 2020-12-17 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumors; Solid Tumors; Ovarian Cancer; Breast Cancer; Prostate Cancer; NSCLC; Pancreatic Cancer; Colorectal Cancer
Keywords: PARP inhibitor; Talazoparib; Talzenna; BRCA mutation; ATM mutation; Pharmacokinetics; Bioequivalence; Bioavailability; Food effect
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms | interventions — talazoparib

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 2 sequences to receive Treatment A, B and C in different order as shown below. The first 2 periods will be for BE assessment, with the first period being 28 days and the following periods being 21 days. Period 3 will be a 21 day period to evaluate the food effect on the PK of the proposed talazoparib soft gel capsule formulation that will be included in the fixed sequence after the 2 BE assessment periods (for participants who can tolerate one high-fat/high-calorie meal). Participants must have received 21 consecutive days of continuous 1mg QD drug administration to be considered as completers of a treatment period, before moving on to the next scheduled treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequence 1 (Experimental): Participants receive Treatment B for 28 days, followed by Treatment A for 21 days, followed by Treatment C for 21 days.
  Interventions: Drug: TALZENNA capsule; Drug: Talazoparib soft gel capsule
- Sequence 2 (Experimental): Participants receive Treatment A for 28 days, followed by Treatment B for 21 days, followed by Treatment C for 21 days.
  Interventions: Drug: TALZENNA capsule; Drug: Talazoparib soft gel capsule

INTERVENTIONS:
Drug: TALZENNA capsule — Current commercial talazoparib formulation 1 mg once daily given under fasting condition
Drug: Talazoparib soft gel capsule — Proposed talazoparib soft gel capsule formulation 1 mg once daily under fasting condition
Drug: Talazoparib soft gel capsule — Proposed talazoparib soft gel capsule formulation 1 mg once daily under fed condition

SUMMARY:
This will be a Phase 1, open label, 2-sequence, crossover study to establish the BE of the current commercial formulation (Generation 3.1 talazoparib capsules) to the proposed talazoparib liquid-filled soft gelatin capsule (soft gel capsule) formulation after multiple dosing under fasting conditions in participants with advanced solid tumors. In addition, the effect of food on the PK of the proposed talazoparib soft gel capsule formulation will be evaluated in fixed sequence after the 2 BE assessment periods.

ELIGIBILITY:
Inclusion Criteria

1. Histological diagnosis of recurrent, locally advanced or metastatic solid tumor that is not amenable for treatment with curative intent.

   * Solid tumors with known or likely pathogenic germline or somatic tumor gene defect (eg, one or more BRCA1 or BRCA2 gene defect except for ovarian cancer) that would benefit from PARPi therapy per current approvals for the tumor indication or supported by strong scientific evidence.
   * Received at least 1 prior SOC regimen, if it exists, as appropriate for the respective tumor type unless deemed unsuitable or declined these therapies; ovarian cancer participants must have at least 1 prior cytotoxic chemotherapy regimen, including at least 1 course of platinum-based therapy. Participants must not have had disease progression within 6 months of initiation of platinum containing regimen.
2. ECOG performance score of 0-1.
3. Adequate bone marrow function:

   * ANC ≥1500 cells/mm3
   * Platelets ≥100,000 cells/mm3
   * Hemoglobin ≥10.0 g/dL
4. Adequate organ functions:

   * CLCR ≥60 mL/min and no documented CLCR <60 mL/min and no change in CLCR >25% in the past 4 weeks
   * AST and ALT ≤2.5 × ULN; if liver function abnormalities are due to hepatic metastasis, then AST and ALT ≤5 × ULN;
   * Total bilirubin ≤1.5 × ULN (≤3 × ULN for Gilbert's syndrome);

Exclusion Criteria

1. For ovarian participants: Non-epithelial tumors or ovarian tumors with low malignant potential (ie, borderline tumors) or mucinous tumors.
2. Toxicities from previous anti-cancer therapies must be resolved to NCI CTCAE <Grade 2, except for alopecia, sensory neuropathies ≤Grade 2, or other Grade ≤2 AEs not constituting a safety risk, based on investigator's judgment, are acceptable.
3. Diagnosed with MDS or AML.
4. Active infection requiring systemic therapy within 2 weeks of enrollment.
5. Any condition in which active bleeding or pathological conditions may carry a high risk of bleeding (eg, known bleeding disorder, coagulopathy or tumor involvement with major vessels).
6. Known or suspected brain metastasis or active leptomeningeal disease undergoing or requiring treatment. Asymptomatic brain metastases currently not undergoing treatment are allowed.
7. Known history of testing positive for HIV, AIDS, positive HBV surface antigen, positive HCV RNA, or positive COVID-19 viral test. Asymptomatic patients with no active infection detected but positive antibody tests, indicating past infection, are allowed.
8. Current or anticipated use of P-gp inhibitors, BCRP inhibitors, and P-gp inducers within 2 weeks or 5 half-lives prior to randomization (whichever is longer) .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (23):
  - California Cancer Associates for Research and Excellence, Inc (cCARE), Encinitas, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Cancer Associates for Research and Excellence, Inc (cCARE), San Marcos, California
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - Florida Cancer Specialists, Lake Mary, Florida
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - NYU Langone Hospital - Long Island Oncology, Mineola, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Investigational Pharmacy, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - West Chester Hospital, West Chester, Ohio
  - UPCI Investigational Drug Service, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Upmc Shadyside, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research - Medical City Hospital, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas
- Australia (8):
  - Liverpool Cancer Therapy Centre, Liverpool, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Monash Health, Clayton, Victoria
  - Epworth Healthcare (Epworth Freemasons Hospital), East Melbourne, Victoria
  - Epworth Healthcare, East Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Epworth Richmond Hospital (Epworth Healthcare), Richmond, Victoria
  - Epworth Healthcare, East Melbourne

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang D, Guo CC, Gao X, Wang Y, Yu Y, Plotka A, Elmeliegy M, Shi H, Johnson S, DeAnnuntis L, Hoffman J. Talazoparib Formulation Bridging in Cancer Patients-Challenges and the Critical Role of Model-Informed Drug Development in Approval Despite Failed Bioequivalence. CPT Pharmacometrics Syst Pharmacol. 2025 Dec 11. doi: 10.1002/psp4.70157. Online ahead of print. PMID 41379622
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 73 participants were assigned to study treatment, and all of them were permanently discontinued from study treatment. Fifty-two participants entered the safety follow-up phase and 46 of them completed the safety follow-up.
Groups:
- Sequence 1: Participants were randomly assigned to sequence BAC. Participants received treatment B: talazoparib soft gel capsule formulation 1 mg once daily given under fasting condition in Period 1 for 28 days followed by Treatment A: current commercial talazoparib formulation 1 mg once daily given under fasting condition in Period 2 for 21 days. Participants received Treatment C: talazoparib soft gelatin capsule formulation 1 mg once daily given with food in Period 3 (food effect assessment) for 21 days. Participants who required a dose reduction, had unstable renal function, experienced renal function worsening to moderate/severe renal impairment during the study, or completed the food effect assessment, were enrolled over to the maintenance phase which consisted of repeating 28- day cycles of treatment with the current commercial talazoparib formulation 1 mg once daily.
- Sequence 2: Participants were randomly assigned to sequence ABC. Participants received treatment A: current commercial talazoparib formulation 1 mg once daily given under fasting condition in Period 1 for 28 days followed by Treatment B: talazoparib soft gel capsule formulation 1 mg once daily given under fasting condition in Period 2 for 21 days. Participants received Treatment C: talazoparib soft gelatin capsule formulation 1 mg once daily given with food in Period 3 (food effect assessment) for 21 days. Participants who required a dose reduction, had unstable renal function, experienced renal function worsening to moderate/severe renal impairment during the study, or completed the food effect assessment, were enrolled over to the maintenance phase which consisted of repeating 28- day cycles of treatment with the current commercial talazoparib formulation 1 mg once daily.
Period: Bioequivalence Phase: Period 1 (28 Days)
Arm/Group | Sequence 1 | Sequence 2
Started | 35 | 38
Completed | 28 | 28
Not Completed | 7 | 10
Not completed — Death | 1 | 2
Not completed — Progressive disease | 2 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Global deterioration of health status | 0 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Other | 1 | 0
Period: Bioequivalence Phase: Period 2 (21 Days)
Arm/Group | Sequence 1 | Sequence 2
Started | 27 (One participant did not start period 2.) | 25 (Three participants did not start period 2.)
Completed | 25 | 20
Not Completed | 2 | 5
Not completed — Progressive disease | 1 | 5
Not completed — Withdrawal by Subject | 1 | 0
Period: Food Effect Phase: Period 3 (21 Days)
Arm/Group | Sequence 1 | Sequence 2
Started | 16 (Nine participants did not start period 3.) | 14 (Six participants did not start period 3.)
Completed | 11 | 11
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Progressive disease | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Refused further treatment | 0 | 1
Not completed — Other | 1 | 0
Period: Maintenance Phase: Period 4 (28 Days)
Arm/Group | Sequence 1 | Sequence 2
Started | 21 (Participants who entered maintenance period.) | 20 (Participants who entered maintenance period.)
Completed | 0 | 0
Not Completed | 21 | 20
Not completed — Adverse Event | 1 | 0
Not completed — Progressive disease | 10 | 12
Not completed — Refused further treatment | 1 | 0
Not completed — Other | 9 | 8

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study treatment.
Groups:
- All Participants: Participants were randomly assigned to 1 of 2 sequences to receive treatments A, B and C in different order with 3 periods. The first 2 periods were for BE assessment with treatment A and B (Period 1 was 28 days and Period 2 was 21 days); Period 3 was a 21-day period to evaluate the food effect with treatment C. Sequence 1 (Period 1: Treatment B; Period 2: Treatment A; Period 3: Treatment C); Sequence 2 (Period 1: Treatment A; Period 2: Treatment B; Period 3: Treatment C); Treatment A: current commercial talazoparib formulation 1 mg once daily given under fasting condition (reference for BE evaluation); Treatment B: the proposed talazoparib soft gel capsule formulation 1 mg once daily given under fasting condition (test for BE evaluation, reference for food effect evaluation); Treatment C: the proposed talazoparib soft gelatin capsule formulation 1 mg once daily given with food (on the PK sampling day, high-fat/high-calorie meal was administered in the clinical sites prior to the administration of the proposed talazoparib soft gelatin capsule formulation; test for food-effect evaluation).
Arm/Group | All Participants
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57
  Black or African American | 11
  Asian | 1
  Not reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 24 Hours (AUC24) of Talazoparib After Multiple Dosing Under Fasted Conditions
Description: AUC24 was defined as area under the plasma concentration-time profile from time zero to 24 hours post dose. The geometric coefficient of variation is expressed in percentage. The ratio (Test/Reference) of adjusted means and 90% CI were expressed as percentages.
Time Frame: Serial blood sample (4 mL) each was collected at predose on Day 27 of Period 1 and Day 20 of Periods 2 and predose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, and 24 hours postdose on Day 28 of Period 1 and Day 21 of Period 2 to 3, respectively.
Population: The analysis population was defined as all participants randomized and treated who had primary PK parameter of AUC24 or Cmax in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/millilitre (ng*hr/mL)
Groups:
- Treatment A: Commercial Capsule Fast: Current commercial talazoparib formulation 1 mg once daily was given under fasted conditions (reference for BE evaluation).
- Treatment B: Soft Gel Capsule Fast: The proposed talazoparib soft gelatin capsule formulation 1 mg once daily was given under fasted conditions (test for BE evaluation, reference for food-effect evaluation).
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast
Number analyzed (Participants) | 47 | 40
nanograms*hour/millilitre (ng*hr/mL) | 178.7 (40) | 173.0 (32)
Statistical Analysis 1: Comparison: Treatment A: Commercial Capsule Fast vs Treatment B: Soft Gel Capsule Fast; Treatment A were reference; treatment B were test; Test type: Other; Mixed Models Analysis; Ratio (Test/Reference) of Adjusted Means = 105.16, 90% CI 2-sided [99.00 to 111.70]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Talazoparib After Multiple Dosing Under Fasted Conditions
Description: Cmax was the maximum observed plasma concentration and was directly observed from data. The geometric coefficient of variation was expressed in percentage. The ratio (Test/Reference) of adjusted means and 90% CI were expressed as percentages.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/millilitre (ng/mL)
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast
Number analyzed (Participants) | 47 | 40
nanograms/millilitre (ng/mL) | 14.95 (40) | 19.19 (32)
Statistical Analysis 1: Comparison: Treatment A: Commercial Capsule Fast vs Treatment B: Soft Gel Capsule Fast; Treatment A were reference; treatment B were test; Test type: Other; Mixed Models Analysis; Ratio (Test/Reference) of Adjusted Means = 136.62, 90% CI 2-sided [125.05 to 149.27]

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 24 Hours (AUC24) of Talazoparib After Multiple Dosing Under Fed Conditions
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Treatment C: Soft Gel Capsule Fed: The proposed talazoparib soft gelatin capsule formulation 1 mg once daily was given with food (on the PK sampling day, high-fat/high-calorie meal was administered in the clinical sites prior to the administration of the proposed talazoparib soft gelatin capsule formulation; test for food-effect evaluation).
Arm/Group | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed
Number analyzed (Participants) | 40 | 21
ng*hr/mL | 173.0 (32) | 151.3 (38)
Statistical Analysis 1: Comparison: Treatment B: Soft Gel Capsule Fast vs Treatment C: Soft Gel Capsule Fed; Treatment B were reference; treatment C were test; Test type: Other; Mixed Models Analysis; Ratio (Test/Reference) of Adjusted Means = 87.97, 90% CI 2-sided [81.82 to 94.58]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Talazoparib After Multiple Dosing Under Fed Conditions
Description: as for outcome 2
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants randomized and treated who had primary PK parameter of AUC24 or Cmax in at least 1 treatment period. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed
Number analyzed (Participants) | 40 | 22
ng/mL | 19.19 (32) | 11.36 (38)
Statistical Analysis 1: Comparison: Treatment B: Soft Gel Capsule Fast vs Treatment C: Soft Gel Capsule Fed; Treatment B were reference; treatment C were test; Test type: Other; Mixed Models Analysis; Ratio (Test/Reference) of Adjusted Means = 58.26, 90% CI 2-sided [51.55 to 65.84]

5. Secondary Outcome: Apparent Clearance After Oral Dose (CL/F) of Talazoparib After Multiple Dosing
Description: Apparent Clearance After Oral Dose (CL/F) was defined as apparent clearance after oral dose on the last day of treatment period. The geometric coefficient of variation is expressed in percentage.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed
Number analyzed (Participants) | 47 | 40 | 21
liter per hour (L/hr) | 5.631 (40) | 5.808 (32) | 6.648 (38)

6. Secondary Outcome: Time of Observed Maximum Plasma Concentration (Tmax) of Talazoparib After Multiple Dosing
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed
Number analyzed (Participants) | 47 | 40 | 22
hour | 2.00 [0.500 to 6.00] | 0.975 [0.417 to 4.00] | 4.00 [0.967 to 24.7]

7. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to Time of the Last Quantifiable Concentration (AUClast) of Talazoparib After Multiple Dosing
Description: AUClast was area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration. The geometric coefficient of variation was expressed in percentage.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed
Number analyzed (Participants) | 47 | 40 | 21
ng*hr/mL | 178.5 (41) | 173.4 (33) | 152.1 (38)

8. Secondary Outcome: Predose Concentration During Multiple Dosing (Ctrough) of Talazoparib After Multiple Dosing
Description: Ctrough was the pre-dose concentration during multiple dosing and was directly observed from data. The geometric coefficient of variation is expressed in percentage.
Time Frame: Serial blood sample (4 mL) each was collected at predose on Day 27 of Period 1 and Day 20 of Periods 2, predose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, and 24 hours postdose on Day 28 of Period 1 and Day 21 of Period 2 to 3, respectively.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed
Number analyzed (Participants) | 47 | 40 | 22
ng/mL | 4.269 (48) | 3.645 (44) | 3.633 (60)

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (All Causalities)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Treatment-emergent adverse event (TEAE) means event between first dose of study treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of death; inpatient hospitalization; life-threatening experience; disability; congenital anomaly or deemed significant for any other reason.
Time Frame: Day 1 up to 28 days after last dose of study drug (maximum up to 388 days)
Population: Population analysis set included all participants randomly assigned to investigational product (IP) and who took at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Groups:
- Maintenance: Participants who had repeated a period 2 times but still could not meet PK evaluable criteria, needed a dose reduction, had unstable renal function, had experienced renal function worsening to moderate/severe renal impairment during the study, or had completed the food effect assessment, was rolled over to the maintenance phase which consisted of repeating 28 day cycles of treatment with the current commercial formulation.
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed | Maintenance
Number analyzed (Participants) | 65 | 60 | 30 | 41
Participants
  Participants with adverse events | 42 | 36 | 15 | 31
  Participants with serious adverse events | 9 | 7 | 1 | 7
  Participants with Maximum Grade 3 or 4 adverse events | 13 | 10 | 5 | 12
  Participants with Maximum Grade 5 adverse events | 3 | 4 | 0 | 1
  Participants discontinued study drug due to adverse events | 3 | 4 | 1 | 2
  Participants with dose reduced or temporary discontinuation due to adverse events | 13 | 9 | 6 | 13

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (Treatment Related)
Description: as for outcome 9
Time Frame: Day 1 up to 28 days after last dose of study drug (maximum up to 388 days)
Population: Population analysis set included all participants randomly assigned to IP and who took at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed | Maintenance
Number analyzed (Participants) | 65 | 60 | 30 | 41
Participants
  Participants with adverse events | 22 | 26 | 11 | 16
  Participants with serious adverse events | 2 | 0 | 0 | 3
  Participants with Maximum Grade 3 or 4 adverse events | 9 | 8 | 4 | 10
  Participants discontinued study drug due to adverse events | 1 | 1 | 0 | 1
  Participants with dose reduced or temporary discontinuation due to adverse events | 9 | 7 | 6 | 12

ADVERSE EVENTS:
Time Frame: From day 1 up to maximum 388 days.
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Treatment A: Commercial Capsule Fast | Treatment B: Soft Gel Capsule Fast | Treatment C: Soft Gel Capsule Fed | Maintenance
All-Cause Mortality (participants affected / at risk) | 4/65 | 5/60 | 0/30 | 1/41
Serious Adverse Events (participants affected / at risk) | 9/65 | 7/60 | 1/30 | 7/41
Other Adverse Events (participants affected / at risk) | 25/65 | 25/60 | 12/30 | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Commercial Capsule Fast (N=65) | Treatment B: Soft Gel Capsule Fast (N=60) | Treatment C: Soft Gel Capsule Fed (N=30) | Maintenance (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Disease progression (General disorders) | 2 | 3 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Commercial Capsule Fast (N=65) | Treatment B: Soft Gel Capsule Fast (N=60) | Treatment C: Soft Gel Capsule Fed (N=30) | Maintenance (N=41)
Anaemia (Blood and lymphatic system disorders) | 7 | 8 | 5 | 11
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 1 | 3
Nausea (Gastrointestinal disorders) | 7 | 5 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 2
Fatigue (General disorders) | 4 | 11 | 2 | 7
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 0 | 0
Platelet count decreased (Investigations) | 4 | 4 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Hypotension (Vascular disorders) | 1 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT04672460/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT04672460/SAP_001.pdf